CLINICAL TRIAL: NCT01878383
Title: Device Trial: Identification of Herpes Simplex Virus (HSV) Shedding in the Female Genital Tract of Pregnant and Nonpregnant Women by GeneXpert PCR, Routine PCR, and Culture
Brief Title: Identification of Herpes Simplex Virus (HSV) Shedding in the Female Genital Tract of Pregnant and Nonpregnant Women by GeneXpert PCR, Routine PCR, and Culture
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Kimberlin, MD, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: DMID 11-0070
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Herpes Simplex Virus
Keywords: (HSV)
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non-pregnant women/active HSV lesions: Women presenting to local health department
  Interventions: Device: Genexpert assay
- Pregnant women/no active HSV lesions: Women presenting in active labor
  Interventions: Device: Genexpert assay

INTERVENTIONS:
Device: Genexpert assay

SUMMARY:
PCR detection of HSV DNA shedding in the female genital tract using the GeneXpert system (Cepheid, Sunnyvale CA) will be compared with traditional (routine) PCR (pregnant and nonpregnant women) and with HSV culture (nonpregnant women). The GeneXpert system performs all sample-processing steps and real-time PCR in a single integrated cartridge. The standard cartridge is an inexpensive disposable plastic cartridge with filtration and ultrasonic lysis capabilities. It consists chiefly of several combined molded plastic components: a cartridge body containing eleven fluid reservoirs or chambers along with an attached PCR tube, a specialized valve body with an ultrasonic interface containing a sub-micron filter and glass lysis beads, and a rotary valve with an axial syringe barrel. The operation of the cartridge is simple. The rotary valve contains an inlet and an outlet port. Fluid such as a sample buffer can be drawn up into a syringe drive through the inlet port of the rotary valve and then dispensed into any other chamber within the cartridge by rotating the valve and expelling the fluid through the outlet port. The fluid can either be passed through a filter contained within the valve assembly or it can be passed directly into the next chamber without filtration, depending on the path that is chosen. The cartridge fluidics and subsequent real-time PCR all are performed within the GeneXpert instrument. The GeneXpert contains multiple modules (ICORE units) that can be independently programmed to drive the syringe/rotary valve, and to perform four-color real-time PCR. Each cartridge fits inside one module, and all processing, PCR, and analysis steps are performed automatically. Each ICORE module can be run and analyzed independently, so batching of samples is unnecessary.

DETAILED DESCRIPTION:
The GeneXpert HSV PCR test will be validated against HSV viral cultures and routine quantitative PCR. Validation will occur in two populations: 1) nonpregnant women in STI clinics with clinically-apparent HSV lesions (Group 1, n=300), and 2) pregnant women in active labor with no visible evidence of HSV infection (Group 2, n=12,500). All testing of samples on the GeneXpert platform, routine quantitative PCR, and viral culture will be done at the UAB Central Laboratory. Women in each group will have specimens obtained from genital lesions (Group 1) or vaginal swabs (Group 2). Specimens from all women in Group 1 will be evaluated by HSV culture, routine HSV PCR, and GeneXpert HSV PCR. Approximately half of the women in Group 2 will be tested by routine HSV PCR and GeneXpert HSV PCR; specimens from the rest of the women in Group 2 will be stored for possible testing in the future by routine HSV PCR and GeneXpert HSV PCR. In this manner, we will maximize the data from which to compare GeneXpert PCR results with routine PCR, while maintaining flexibility to ensure an adequate number of specimens are positive for HSV DNA by routine PCR.

Swabs from pregnant women in labor will be placed in viral transport media, frozen at -20°C, and batch-shipped to the UAB Central Laboratory for analysis on the GeneXpert instrument and by routine HSV quantitative PCR. Swabs from nonpregnant women in STI clinics will be placed in viral transport media, refrigerated at 4°C, and shipped to the UAB Central Laboratory for real time analysis on the GeneXpert instrument and by HSV culture and routine quantitative HSV PCR. Specimens from the first 300 women enrolled in Group 2 will be run as individual routine PCRs and in batches of 5 samples per PCR run. In this manner, we will validate that the level of detection from batching of samples for routine PCR is acceptable. Once this validation occurs, specimens from the approximately half of remaining Group 2 women will be batched for real-time routine PCR analysis. If a batch run of 5 specimens is negative, no further testing will be performed. If a batch run of 5 specimens is positive, all of the specimens will be separated out for re-running as individual PCRs. All specimens evaluated by routine PCR will also be evaluated by GeneXpert PCR; in this manner, we will have individual routine PCR results results for comparison against GeneXpert PCR results.

A blood specimen will be obtained from each nonpregnant (Group 1) and pregnant (Group 2) woman at the time of enrollment, and if she is determined to be shedding HSV by routine PCR, GeneXpert PCR, or culture then type-specific serologic testing will be performed. Correlation of viral typing from the virologic sampling with HSV-1 and HSV-2 serostatus will allow for categorization of infection (first-episode primary, first-episode nonprimary, or recurrent infection).

Those women in Group 1 who have a positive HSV culture will be contacted directly when the result is known. Women in Group 2 with a positive HSV PCR result will not be contacted because routine HSV PCR and GeneXpert PCR are not FDA-cleared tests in this population; thus, we will not know the test performance characteristics (e.g., sensitivity, specificity, etc.) until completion of the trial. All pregnant women in Group 2 will receive written materials at the time of enrollment educating them on signs and symptoms of neonatal HSV disease. All postpartum women will be contacted by telephone 60-90 days post-delivery and an inquiry will be made to determine if their babies developed neonatal HSV disease.

Data on the incidence of neonatal HSV disease among babies delivered to women in Group 2 will be compared with the incidence data from Brown et al.1 In their study of almost 60,000 women conducted over a 20 year period, this group of researchers has reported an incidence rate for neonatal HSV disease of 1 in 3,200 live births.

ELIGIBILITY:
Inclusion Criteria:•Signed Informed Consent from woman

•≥ 19 years of age

* Female gender
* In active labor with a viable fetus, OR non-pregnant and being evaluated in STI clinics for herpetic genital lesions

Exclusion Criteria:•For women in active labor, active herpetic lesions in the genital region

* Receipt of acyclovir, valacyclovir, or famciclovir within the previous 14 days
* Known HIV infection

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant and non-pregnant women
Sampling Method: Probability Sample
Enrollment: 12550 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Kimberlin, MD, Principal Investigator — University of Alabama at Birmingham; Richard Whitley, MD, Principal Investigator — University of Alabama at Birmingham
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Colorado at Denver Health Sciences Center, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory Children's Center, Atlanta, Georgia
  - Louisiana State University Health Science Center-Shreveport, Shreveport, Louisiana
  - Washington University in St Louis School of Medicine, St Louis, Missouri
  - Dartmouth Medical School, Lebanon, New Hampshire
  - Steven & Alexandra Cohen Children's Medical Center of New York (CCMC), Manhasset, New York
  - University of Rochester Medical Center, Rochester, New York
  - Carolinas Medical Center - Charlotte, Charlotte, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Nationwide Children Hospital, Columbus, Ohio
  - McGee Women's Hospital, Pittsburgh, Pennsylvania
  - University of Utah School of Medicine, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-pregnant Women/Active HSV Lesions: Women presenting to local health department
  Genexpert assay
- Pregnant Women/no Active HSV Lesions: Women presenting in active labor will be tested for HSV utilizing the Genexpert assay
Period: Overall Study
Arm/Group | Non-pregnant Women/Active HSV Lesions | Pregnant Women/no Active HSV Lesions
Started | 50 | 12500
Completed | 50 | 11001
Not Completed | 0 | 1499
Not completed — Lost to Follow-up | 0 | 1499

BASELINE CHARACTERISTICS:
Groups:
- Pregnant Women/no Active HSV Lesions: Women presenting in active labor
  Genexpert assay
- Total: Total of all reporting groups
Arm/Group | Non-pregnant Women/Active HSV Lesions | Pregnant Women/no Active HSV Lesions | Total
Number analyzed (Participants) | 50 | 12500 | 12550
Age, Continuous [Median (Standard Deviation); unit: Years] — Age was not collected Population: Age was not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 12500 | 12550
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline information not available for 2 subjects
  Participants
    number analyzed (Participants) | 50 | 12498 | 12548
    Hispanic or Latino | 1 | 1090 | 1091
    Not Hispanic or Latino | 49 | 11124 | 11173
    Unknown or Not Reported | 0 | 284 | 284
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographic information not available for 2 subjects.
  Participants
    number analyzed (Participants) | 50 | 12498 | 12548
    American Indian or Alaska Native | 0 | 39 | 39
    Asian | 0 | 335 | 335
    Native Hawaiian or Other Pacific Islander | 0 | 23 | 23
    Black or African American | 43 | 4631 | 4674
    White | 7 | 6859 | 6866
    More than one race | 0 | 225 | 225
    Unknown or Not Reported | 0 | 386 | 386

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Detection of HSV DNA by GeneXpert PCR From Specimens Obtained From the Genital Tract of Non-pregnant Women in STI Clinics, as Compared With HSV Culture
Description: Assessing the vaginal specimen collected via a swab of non-pregnant women presenting to their provider at the time of active HSV outbreak with standard HSV culture compared to the assay of new device called a GeneXpert.
  Percent of GeneXpert assessment in agreement with standard HSV culture, for subjects who were positive for HSV according to culture.
Time Frame: on day of enrollment
Measure: Number (95% Confidence Interval); unit: Sensitivity (percent positive)
Arm/Group | Non-pregnant Women/Active HSV Lesions
Number analyzed (Participants) | 50
Sensitivity (percent positive) | 100 [90.8 to 100]
Statistical Analysis 1: Comparison: Non-pregnant Women/Active HSV Lesions; Test type: Other — Sensitivity is the percent of non-pregnant women positive for shedding HSV by culture method in which GeneXpert test results is positive. Units equals percent non-pregnant women positive; Sensitivity = 100, 95% CI 2-sided [90.8 to 100] — 95% Clopper-Pearson Exact Confidence Interval

2. Primary Outcome: Positive Percent Agreement of Detection of HSV DNA by GeneXpert PCR From Specimens Obtained From Genital Tract of Pregnant Women, as Compared With Routine PCR Detection of Viral DNA
Description: Detection of HSV DNA by GeneXpert PCR compared to routine PCR detection by viral DNA. Percent of GeneXpert assessment in agreement with routine PCR detection, for subjects who are positive for HSV according to routine PCR.
Time Frame: DAY OF ENROLLMENT
Population: 12,500 pregnant women were enrolled into this study and were randomized (1:1) to either have their specimens stored or tested. The analysis population is the 6,658 subjects randomized to the test condition
Measure: Number (95% Confidence Interval); unit: Positive percent agreement
Arm/Group | Pregnant Women/no Active HSV Lesions
Number analyzed (Participants) | 6658
Positive percent agreement | 80 [73.7 to 86.3]
Statistical Analysis 1: Comparison: Pregnant Women/no Active HSV Lesions; Test type: Other — Positive percent agreement is the percent of pregnant women with positive routine PCR results in which GeneXpert test results is positive. Units equal percent of pregnant women positive; Positive percent agreement = 80, 95% CI 2-sided [73.7 to 86.3] — 95% large sample confidence interval

3. Primary Outcome: Negative Percent Agreement of Detection of HSV DNA by GeneXpert PCR From Specimens Obtained From Genital Tract of Pregnant Women, as Compared With Routine PCR Detection of Viral DNA
Description: Detection of HSV DNA by GeneXpert PCR compared to routine PCR detection by viral DNA. Percent of GeneXpert assessments in agreement with routine PCR detection, for subjects who were negative for HSV according to routine PCR.
Time Frame: DAY OF ENROLLMENT
Population: 12,500 pregnant women were enrolled into this study and were randomized (1:1) to either have the specimens stored or tested. The analysis population is the 6,658 subjects randomized to the test condition
Measure: Number (95% Confidence Interval); unit: Negative percent agreement
Arm/Group | Pregnant Women/no Active HSV Lesions
Number analyzed (Participants) | 6658
Negative percent agreement | 99.2 [99 to 99.5]
Statistical Analysis 1: Comparison: Pregnant Women/no Active HSV Lesions; Test type: Other — Negative percent agreement is the percent of pregnant women with negative routine PCR results in which GeneXpert test results is negative. Units equal percent of pregnant women negative; Negative percent agreement = 99.2, 95% CI 2-sided [99 to 99.5] — 95% large sample confidence interval

ADVERSE EVENTS:
Time Frame: 1 day for group 1 (non-pregnant); 30-90 for group 2 (pregnant)
Description: No adverse events were reported
Arm/Group | Non-pregnant Women/Active HSV Lesions | Pregnant Women/no Active HSV Lesions
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/12500
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/12500
Other Adverse Events (participants affected / at risk) | 0/50 | 0/12500

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT01878383/Prot_SAP_000.pdf